CLINICAL TRIAL: NCT06511323
Title: Evaluation of Brain Metastases Treated With Stereotactic Radiotherapy Using Dynamic [18F]FDG PET
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Melody Qu, Radiation Oncologist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 124854
Record Dates: First submitted 2024-06-27; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Brain Metastases
Keywords: Dynamic F-18 FDG PET,; Brain metastases; Stereotactic radiation; Radio-necrosis; Pseudo-progression
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Observational (Experimental): This is a prospective, single-arm, pilot diagnostic study to evaluate the diagnostic accuracy of using dynamic [18F]FDG PET in 70 patients with brain metastases managed with stereotactic radiosurgery(SRS)/fractionated stereotactic radiotherapy (FSRT). The study will include imaging assessments at baseline, at 10 weeks after treatment, and at first concern for progression or 12 months post-treatment, whichever comes earlier.
  Interventions: Diagnostic Test: dynamic [18-FDG PET] scan post stereotactic radiation for brain metastases

INTERVENTIONS:
Diagnostic Test: dynamic [18-FDG PET] scan post stereotactic radiation for brain metastases — at baseline prior to stereotactic radiation, at 10 weeks after treatment, and at first concern for progression at treated lesion or 12 months post-treatment, whichever comes earlier.

SUMMARY:
The purpose of this study is to evaluate the clinical usefulness of dynamic [18F]FDG PET imaging in assessing brain metastasis post stereotactic radiotherapy to separate true progression from the treatment-related changes.

DETAILED DESCRIPTION:
After being informed about the study and potential risk, all participants giving written informed consent will be screened to determine if participant being referred fits eligibility criteria for the study, under of the supervision of the radiation oncologist. If a participant agrees to participate in this study, they will receive three additional imaging sessions (the dynamic PET scan). The first session will occur prior to starting treatment; the second session will occur at about 10 weeks post treatment; the third session will occur at first concern of progression at treated lesions or 12 months post-treatment, whichever comes earlier. These scans will be scheduled in addition to the participant's regular follow-up scans and appointments.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older.
* Willing and able to provide consent.
* ECOG 0-2.
* Life expectancy ≥12 months.
* Creatinine clearance ≥30 ml/min within 28 days prior to registration.
* At the discretion of the treating oncologist, it is believed that at least 1 lesion (or resection cavity) is best managed with SRS/SFR

Exclusion Criteria:

* Pregnant or nursing women.
* Men or women of childbearing potential who are unwilling to employ adequate contraception.
* Inability to complete a brain MRI.
* Known allergy to gadolinium.
* Inability to complete a PET scan.
* Uncontrolled diabetes mellitus.
* Primary germ cell tumour, primary CNS tumour, or lymphoma
* SRS/FSRT is no longer indicated for any BMs
* Must be able to read and write English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of dynamic PET | 12-month follow-up.
  Diagnostic accuracy will be calculated and compared based on the index lesion.

SECONDARY OUTCOMES:
Clinical outcomes | 24-month follow-up
  Clinical outcomes such as local recurrence.
Clinical outcomes | 24-month follow-up
  CNS progression-free survival and overall survival will be analyzed
Clinical outcomes | 24-month follow-up
  Factors impact on these outcomes will be explored.
Diagnostic imaging outcomes | 24-month follow-up
  GMR-to-perfusion ratio.
Diagnostic imaging outcomes | 24-month follow-up
  Blood-brain barrier permeability to glucose.
Diagnostic imaging outcomes | 24-month follow-up
  Glucose Metabolic Rate.
Diagnostic imaging outcomes | 24-month follow-up
  Magnetic resonance spectroscopy data.
Diagnostic imaging outcomes | 24-month follow-up
  Other ancillary clinical data will be explored.
Cost-effectiveness analysis | 24-month follow-up
  A decision analysis model coupled with Markov model will be constructed to estimate the incremental cost-effectiveness ratio (ICER) of performing dynamic PET in this setting from the Canadian health-care system perspective.

IPD SHARING:
Plan to Share IPD: No